CLINICAL TRIAL: NCT00002299
Title: Combination Therapy With 9-(1,3-Dihydroxy-2-Propoxymethyl) Guanine (DHPG) and Interferon Beta for the Prevention of Relapse of Cytomegalovirus Retinitis in Patients With the Acquired Immunodeficiency Syndrome
Brief Title: The Safety and Effectiveness of Ganciclovir Plus Interferon Beta in Preventing the Return of Cytomegalovirus (CMV) of the Eyes in Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 017A; ICM 1285
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-04

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; AIDS-Related Opportunistic Infections; Ganciclovir; Drug Therapy, Combination; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome; Interferon Type I
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; AIDS-Related Opportunistic Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Interferon beta-1b; Ganciclovir

INTERVENTIONS:
Drug: Interferon beta-1b
Drug: Ganciclovir

SUMMARY:
The use of ganciclovir (DHPG) in combination with interferon beta to prevent relapse of cytomegalovirus retinitis in patients with AIDS. While early clinical trials have shown that 30 mg/kg/week of DHPG is usually sufficient to delay or prevent relapse, neutropenia is a common dose-limiting problem in about 50 percent of patients. Since in vitro data have suggested that there is synergism between DHPG and interferon beta against cytomegalovirus, a reduced dose of DHPG in combination with a low dose of interferon beta may prevent relapse without causing neutropenia. If remission can be maintained with low-dose DHPG and interferon beta, maintenance therapy with a moderate dose of interferon beta alone will be evaluated in a subsequent protocol.

ELIGIBILITY:
Inclusion Criteria

Patients must fulfill the CDC criteria for the diagnosis of AIDS. In addition, patients must have a typical clinical picture of cytomegalovirus (CMV) retinitis, a positive CMV culture from any site, and no other possible explanation for the retinal findings (e.g., toxoplasmosis infection). Patients with AIDS in whom CMV retinitis is suspected will be examined by an ophthalmologist and, if, retinal lesions are seen, shall have a complete set of retinal photographs taken. CMV cultures of throat, buffy coat, urine, and if possible, semen will be obtained.

* Cytomegalovirus and toxoplasmosis serologic (IgG and IgM) tests will also be performed.

Exclusion Criteria

Co-existing Condition:

Patients not meeting inclusion criteria are excluded.

Patients not meeting inclusion criteria are excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - USC, Los Angeles, California
  - UCI Med Ctr, Orange, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Stanford Univ School of Medicine, Stanford, California
  - Univ TX Galveston Med Branch, Galveston, Texas